CLINICAL TRIAL: NCT07094997
Title: Effectiveness of Massage Therapy Among Healthcare Workers Suffering From Low Back Pain - a Randomized Controlled Trial
Brief Title: Massage Therapy for Healthcare Staff
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Kassolik, Phd, PhD, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Massage for healthcare staff
Record Dates: First submitted 2025-07-29; First posted 2025-07-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
Keywords: Randomiezed controlled trial; Massage therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective, three-arm, parallel-group, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guideline-Based Massage Therapy + Self-Massage Group (GMT+SM) (Experimental): GMT+SM - Massage protocol based on guidelines from the Polish Society of Physiotherapy, the Polish Society of Family Medicine, the College of Family Physicians in Poland, and the European Rural and Isolated Practitioners. Delivered by licensed therapists.
  Self-Massage Training:
  One in-person instructional session, plus take-home materials (videos and printed instructions).
  Interventions: Other: Guidline-basaed massage therapy
- Guideline-Based Massage Therapy (GMT) (Experimental): GMT - Massage protocol based on guidelines from the Polish Society of Physiotherapy, the Polish Society of Family Medicine, the College of Family Physicians in Poland, and the European Rural and Isolated Practitioners. Delivered by licensed therapists.
  Interventions: Other: Guidline-basaed massage therapy
- Control group (CG) (Active Comparator): Participants receive Swedish massage
  Interventions: Other: Swedish massage

INTERVENTIONS:
Other: Guidline-basaed massage therapy — Massage protocol based on guidelines from the Polish Society of Physiotherapy, the Polish Society of Family Medicine, the College of Family Physicians in Poland, and the European Rural and Isolated Practitioners
  Arms: Guideline-Based Massage Therapy (GMT); Guideline-Based Massage Therapy + Self-Massage Group (GMT+SM)
Other: Swedish massage — A classical form of therapeutic massage that uses a combination of long, flowing strokes, kneading, friction, tapping, and gentle stretching to promote relaxation, improve circulation, and reduce muscle tension. It is typically performed using oil or lotion to reduce friction on the skin. Techniques are applied with light to moderate pressure and are designed to enhance general well-being and support recovery from muscular discomfort or stress
  Arms: Control group (CG)

SUMMARY:
The piriformis muscle can be a contributing factor to low back pain (LBP) due to its anatomical proximity to the sciatic nerve and sacroiliac joint. When the piriformis becomes tight or irritated, it may compress or irritate the sciatic nerve-a condition often referred to as piriformis syndrome-leading to pain that radiates from the lower back to the buttock and down the leg.

The goal of this clinical trial is to examine the effectiveness of massage therapy in counteracting symptoms of low back pain (LBP) among healthcare workers. The main question it aims to answer is:

- Can massage of the piriformis muscle and related musculature effectively reduce symptoms in individuals experiencing LBP linked to myofascial or neuromuscular dysfunction?

Massage therapy targeting the piriformis and associated muscles (e.g., gluteus maximus, medius, and deep hip rotators) can help by:

* Reducing muscle tension and spasms,
* Improving local blood circulation,
* Alleviating pressure on the sciatic nerve,
* Restoring hip mobility and muscle balance.

DETAILED DESCRIPTION:
Background and Rationale Low back pain (LBP) is a prevalent musculoskeletal condition, particularly among healthcare workers due to occupational stress and physical demands. The piriformis muscle, located in the deep gluteal region, plays a crucial role in hip stabilization and external rotation. Due to its anatomical proximity to the sciatic nerve and sacroiliac joint, hypertonicity or irritation of the piriformis muscle may lead to compression of the sciatic nerve-a condition clinically recognized as piriformis syndrome-which manifests as radiating pain from the lower back through the buttock and into the posterior thigh and leg.

Myofascial and neuromuscular dysfunctions of the piriformis and surrounding musculature (including the gluteus maximus, gluteus medius, and deep lateral rotators) are increasingly implicated in chronic, nonspecific LBP. Massage therapy interventions targeting these soft tissue structures may reduce neuromuscular hyperactivity, restore muscular balance, and decrease nociceptive input. However, there is limited high-quality evidence evaluating the comparative effectiveness of professional massage therapy alone versus in combination with self-massage techniques for addressing piriformis-related LBP.

Additionally, there is no standardized approach based on guidelines developed by medical associations. There is a clear need to formulate and evaluate evidence-based protocols for the management of low back pain (LBP). This study will focus on implementing and assessing guidelines provided by the Polish Society of Physiotherapy, the Polish Society of Family Medicine, and European rural health organizations.

Techniques used during the intervention include targeted soft tissue mobilization focused on:

* Piriformis
* Gluteus maximus and medius
* Obturator internus/externus
* Quadratus femoris

Introducing self-massage as a complementary component to professional massage therapy is essential for sustaining and enhancing therapeutic outcomes in the management of low back pain. While manual therapy sessions provide targeted relief by reducing muscle tension, improving circulation, and alleviating nerve compression, these effects can be transient without ongoing maintenance. Self-massage empowers patients to actively participate in their own care by enabling regular myofascial release and muscle relaxation outside the clinical setting. This continued intervention helps prevent the recurrence of muscle tightness and neuromuscular dysfunction, promotes long-term improvements in tissue flexibility and blood flow, and supports sustained pain reduction and functional restoration. Incorporating self-massage training into treatment protocols fosters patient autonomy, improves adherence to therapy, and ultimately contributes to more durable and meaningful clinical benefits.

In the study researchers try to evaluate the effectiveness of guideline-based massage therapy alone versus guideline-based massage therapy combined with self-massage training, compared to a control group, in improving pain, function, and overall well-being in individuals with a low back pain.

Patients participating in this research on massage and self-massage for low back pain (LBP) can experience several important benefits. Firstly, they may gain access to specialized, guideline-based manual therapy delivered by licensed professionals, which can help reduce pain intensity, relieve muscle tension, and improve mobility in the lower back and hip region. Additionally, those in the self-massage group will acquire practical skills and knowledge to manage their symptoms independently, empowering them with effective techniques to maintain and prolong therapeutic effects between treatment sessions. Participation also offers close monitoring of their condition through regular assessments, which may lead to personalized adjustments in care. Beyond physical improvements, engaging in the study can enhance overall well-being and function, potentially reducing work-related disability and improving quality of life. Finally, contributing to this research advances scientific understanding of effective LBP treatments, potentially benefiting broader patient populations in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthcare workers
* Aged 30-65 years with chronic nonspecific low back pain for ≥3 months
* No medical contraindications to massage therapy
* Body mass index (BMI) between 18.5 and 25 kg/m²
* Provided written informed consent

Exclusion Criteria:

* Massage therapy within the past 3 months
* Contraindications to massage therapy
* Ongoing physical therapy
* Significant medical or psychiatric conditions

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
VAS scale | From enrollment to the end of treatment at 2 weeks
  Visual Analogue Scale (VAS) is a continuous scale consisting of a horizontal line, 100 mm long, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 10). VAS is frequently used to determine the effectiveness of treatment as an outcome measure. Most studies show that VAS is a valid and reliable scale.
ODI | From enrollment to the end of treatment at 2 weeks
  The ODI (Oswestry Disability Index) is a standardized questionnaire used to measure a patient's level of disability due to lower back pain. It assesses how back pain affects a person's ability to manage everyday life.

SECONDARY OUTCOMES:
Thermography | From enrollment to the end of treatment at 2 weeks
  Thermal images taken before and after a massage session can be used to observe temperature changes in specific body areas. An increase in surface temperature is often interpreted as a sign of enhanced blood flow, vasodilation, and localized circulation improvement - all considered typical outcomes of massage.
Doppler USG | From enrollment to the end of treatment at 2 weeks
  Doppler ultrasound is used to assess blood flow in vessels by measuring changes in the frequency of sound waves reflected from moving red blood cells. Velocity and direction of blood flow can be visualized and quantified in real time. Abnormalities such as blockages, narrowing, or turbulence can be detected without the need for invasive procedures. Color and spectral Doppler modes are typically employed to provide detailed flow information. This method is widely considered a reliable, non-invasive tool in vascular diagnostics. In this project arteria glutea superior and inferior will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof K Principal Investigator, Principal Investigator — Department of Massage and Physiotherapy, Wroclaw University of Health and Sport Sciences, Wroclaw, Poland
Locations (1):
- Uniwersytecki Szpital Kliniczny we Wrocławiu, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No